CLINICAL TRIAL: NCT00208572
Title: A Randomized Placebo-Controlled Trial of Citalopram for Anxiety Disorders Following Traumatic Brain Injury
Brief Title: Treatment of Citalopram for Anxiety Disorders Following a Traumatic Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: The Defense and Veterans Brain Injury Center (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); Hunter Holmes McGuire VA Medical Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); 59th Medical Wing (U.S. Federal Agency); James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-71013; WU#03-71013
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-10

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Anxiety Disorders; SRI Treatment
MeSH Terms: conditions — Brain Injuries, Traumatic; Anxiety Disorders | interventions — Citalopram

INTERVENTIONS:
Drug: Citalopram

SUMMARY:
The proposal will assess the effectiveness of SRI treatment of anxiety following TBI. We hypothesize that participants will report significantly fewer and less severe anxiety symptoms after a 12-week course of citalopram than after a 12-week course of placebo.

DETAILED DESCRIPTION:
Anxiety occurs commonly after traumatic brain injury and may influence cognitive, behavioral, and somatic presentations that may interfere with patients' recovery and adaptation to life after brain injury. TBI involves both diffuse brain injury as well as frequent focal injuries to frontal and temporal structures, including hippocampus and amygdala, areas that are also implicated in the neurobiology of anxiety. Although there are anecdotal reports of the benefits of SRIs in the treatment of anxiety in association with TBI, there are unfortunately no controlled trials to establish SRI efficacy in patients whose anxiety is considered secondary to brain injury.

A randomized placebo controlled clinical trial design will be used to investigate the effectiveness of citalopram in patients with anxiety disorder due to a general medical condition, specifically traumatic brain injury (TBI). Beneficiaries who are between 3 and 24 months post injury and who meet criteria for DSM-IV diagnosis of anxiety disorder due to TBI will be recruited from the 7 DVBIC VA and Military Medical Centers. Participants will be randomized to receive an increasing dose of citalopram or placebo up to a dose of 40 mg of citalopram or 4 pills of placebo over a 12-week treatment period. Patients will receive comprehensive multidisciplinary evaluations at a DVBIC site, including neurology, neuropsychology and psychiatry interviews and evaluations at baseline, 12 weeks and 12 months.

Participants will sign informed consent prior to the administration of research tests and scales. An informational script is read to individuals seen within the protocol timeframe. This script will provide a necessary standardization for the presentation of the protocol to potential participants. It also specifies the research coordinator as the individual to present the protocol, rather than a primary clinical care provider. After the script is read, the individual will be given the informed consent to review.

Patients will not be eligible to participate/consent to participate in the study until they reach a Rancho Los Amigos level of 7 or 8. If there is any question as to a patient's capacity to consent, the neuropsychologist and/or psychiatrist involved in the study will assess the subject's intellectual and mental faculties prior to consent. Any confusional state prohibits a subjects from being rated as a 7 or 8. Additionally, in our experience, most patients are not able to undergo a full evaluation in the Walter Reed DVBIC program until they reach this level of recovery. Therefore, we anticipate that almost all patients evaluated in our program will have the capacity to give informed consent.

After signing the volunteer informed consent, the tests and scales will be administered and patients will be randomized to receive a 12-week course of citalopram or placebo. Female participants of childbearing potential will be given a serum pregnancy test (up to 1 tablespoon) prior to being randomized to the study medication. If the result of this test is positive, she will not be allowed to participate in this study. The study physician will discuss alternative treatment options.

Patients will receive an increasing dose of citalopram or placebo up to a dose of 40 mg of citalopram or 4 pills of placebo. See Table 2 for dosing schedule. A blood sample (up to 1 tablespoon) drawn after completion of the 12-week treatment period will be used to obtain citalopram levels as a measure of medication compliance. A two-week taper will follow the treatment period. Patients will receive comprehensive multidisciplinary evaluations at a DVBIC site, including neuropsychological and psychiatric interviews and evaluations at baseline, 12 weeks and 12 months.

Because no randomized, controlled trials exist to suggest that current medical treatment is effective in these patients, and because a substantial placebo effect is a known reality, the design of this study (citalopram vs. placebo) is appropriate. Patients are commonly referred to the DVBIC with mild-moderate mood and anxiety symptoms. We have cared for several clinically anxious patients who refused medications. We worked with them in a supportive educational framework, and in some cases, their anxiety remitted. Thus, the best treatment for these patients is far from established. It is likely that this and other future research will help clarify which treatments are best for which patients.

All patients will be contacted weekly (in person or by phone) during the medication phase to assess general condition, current symptoms and compliance. Female participants will also be asked if there is a possibility that she may be pregnant. If there is a chance, she will be discontinued from the study medication and asked to return to the clinic for a serum pregnancy test. If the result of this test is positive, she will be followed by the study staff for the remainder of the study. If the result of this test is negative, she will be re-started on the study medication at 1 pill or 10 mg of citalopram or placebo per day.

Patients will be rated for improvement at weeks 3, 6, and 9 for possible dosage adjustment. The determination of medication adjustment will be made based upon scores on the Clinical Global Improvement Scale given to the participant at these time points (see Table 2). Dosage adjustment will be considered if the clinician rates the patient as a score of 3 or higher on this scale (Minimally Improved to Very Much Worse). However, the CGI Efficacy Index for drug effect will determine the direction of dosage adjustment. A side effect that is rated as significantly interfering with patient functioning or outweighing therapeutic effect will result in one or more of the following courses of action: (1) addition of concomitant medication, (2) decrease in the study agent dose, (3) discontinuation of the study agent. In other words, a patient who is scored as 3 or higher on the CGI Global Improvement Scale who does not have significant side effects on the CGI Efficacy Index will have the study agent dose increased. Any patient who experiences significant side effects at any time during the treatment period will be considered for dose decrease, discontinuation or concomitant medication use. A decision regarding the proper course of action will be dependent on the severity of the side effect, overall therapeutic effect and patient input.

Patients will return to the study center at the end of the 12-week treatment period for the follow-up evaluation. After the 12-week evaluations, patients will be tapered off citalopram or placebo within 2 weeks. Tapering and discontinuation of the study medication or placebo will be done on a gradual basis (e.g., If the patient is on 30 mg, s/he could take 20 mg for 1 week, 10 mg for one week, then D/C). If, following the 12-week participation in the treatment protocol and the 1-2 week taper period, subjects have recurrent symptoms that are distressing to them or believe they need medication to keep their symptoms from recurring they will be evaluated clinically.

Once participants complete the 12- week treatment period, they will be tapered off the study agent. After the taper has been completed, they may be treated with any therapy or pharmacological intervention that their physician feels is clinically indicated. Although we will be collecting data for one year after participants complete the treatment phase, our primary outcome measures will be collected at the end of the 12th week of the treatment period. We will record all concomitant medications used during the study and all medications being used at the follow-ups for data analysis.

Following the 12-week treatment period and taper, patients may be offered appropriate treatment, including citalopram, if medically indicated. All treatment drugs will be recorded. The blind will not yet be broken, that is, patients will not be able to learn if they were being treated with placebo or citalopram.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury patients between 3 and 24 months post injury.
* Clear evidence/documentation of brain injury:

  i. documented/witnessed loss of consciousness, post traumatic amnesia ii. alteration in mental status (dazed/confused), and/or physical evidence of iii. trauma (MRI/CT hemorrhage/contusion)
* Traumatic brain injury with recovery to a Rancho los Amigos level 7 or 8 (alert and oriented).
* Meet criteria for DSM IV diagnosis Anxiety Disorder Due to a General Medical Condition.
* The symptoms of the anxiety disorder are not being controlled adequately with or without treatment at the time of referral.
* Military or Veteran beneficiary
* Men and non-pregnant/non-breastfeeding females
* Aged 18-65

Exclusion Criteria:

* Severe prior neurologic or psychiatric illness (based on DSM-IV criteria), such as stroke or psychosis. (Previous non-psychotic depression/anxiety is not an exclusion criterion)
* Current/prior unstable medical condition that could affect current brain function (ex. clear anoxic episode, cardiac arrest, current uncontrolled diabetes)
* Contraindication to the use of citalopram.
* Concomitant use of monoamine oxidase inhibitors (MAOIs), cimetidine, lithium, theophylline, digoxin, sumatriptan, warfarin, carbamazepine, triazolam, ketoconazole, CYP3A4 and 2C19 inhibitors, and metoprolol.
* Hypersensitivity to citalopram or any of the inactive ingredients in Celexa®
* Previous severe traumatic brain injury (defined as TBI with period of unconsciousness greater than 1 week. This exclusion refers only to TBIs prior to the current injury.
* Pregnancy (blood test required for females)
* Breastfeeding
* Current active suicidal ideation
* Inability to discontinue other psychotropic medications, such as tricyclic antidepressants or another SRI
* Current drug/alcohol abuse or dependence
* Previous unsuccessful trial of citalopram
* Participation in a concurrent drug or treatment trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2003-11; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
DSM-IV diagnostic criteria for Anxiety Disorder Due to General Medical Condition
Spielberger State Anxiety Inventory

SECONDARY OUTCOMES:
Other psychiatric and psychosocial scales
Neuropsychological test scores
Work Status and Military Duty Status

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jaffee, MD, Principal Investigator — The Defense and Veterans Brain Injury Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States